CLINICAL TRIAL: NCT03277742
Title: Evaluation of an Integral Strategy for Joint Management of DM2 and Pulmonary TB in Orizaba, Veracruz.
Brief Title: Joint Management of DM2 and Pulmonary TB in Orizaba, Veracruz
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to safety reasons. The region was considered too dangerous.
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Guadalupe Delgado Sanchez, Level I National Researchers System, Instituto Nacional de Salud Publica, Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI 1422
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Pulmonary Tuberculosis; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Tuberculosis, Pulmonary; Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): This arm will receive the standard of care for patients with TB and DM2
  Interventions: Drug: Standard of care
- Intervention (Experimental): This arm will receive the community intervention
  Interventions: Behavioral: Community intervention

INTERVENTIONS:
Behavioral: Community intervention — Training of patients, health personnel and community health workers. Bidirectional screening. Monitoring blood glucose levels. Home visits. Medical referral. DOTS.
  Arms: Intervention
Drug: Standard of care — DOTS plus standard DM2 care
  Arms: Control

SUMMARY:
The objective of this study is to evaluate an integral strategy in which diabetes mellitus 2 (DM2) and pulmonary tuberculosis (TB) are managed together. The researchers propose a community intervention with two arms in 4 health centers in Orizaba, Veracruz. Patients will be assigned to either arm by convenience. One arm will receive the joint treatment strategy and another the routine treatment used in health services.

DETAILED DESCRIPTION:
In Mexico DM2 is the main complication of patients with TB (22.2%), more so than HIV, malnutrition and chronic pulmonary obstructive disease (COPD).

The World Health Organization (WHO) has proposed a framework for the joint management of TB and DM2 and one of the key points is the need for studies that evaluate the viability and efficacy of programs that manage both diseases jointly. There are social and clinical determinants that are associated to a higher mortality in patients with DM2 and TB such as poor glucose level control (glycosylated hemoglobin >7mg/dl) and immunosuppression which in turn increases the risk of developing a recurrent episode of TB, being multi drug resistant (MDR) and/or failing TB treatment. The determinants associated to TB are the lack of awareness of the disease, drug toxicity and interaction with DM2 medication and treatment default. Social determinants are low income level, living in a crowded household, living in rural areas, not having access to health care, having been in prison and living with people with TB.

The strategy consists of interventions on patients, health personnel, community health workers and directors of health services. Researchers will train patients in the use of glucometers, health personnel in management of comorbidities of DM2 and TB, health workers in how to support patients and increase treatment adherence. Bidirectional screening in patients with TB or DM2 using bacilloscopies and glycosylated hemoglobin (HbA1c). During the 6 months of directly observed treatment (DOTS) study nurses will monitor levels of glucose weekly with capillary glucose, monthly with fasting glucose, in months 1, 3 and 6 with HbA1c. Patients with high glucose levels will be referred to metabolic control which will be assessed by experts. Regarding DOTs, first line TB drugs will be available and study nurses will supervise that they are taken correctly. A nutritionist will carry out home visits to guide dietary intake.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active PTB, Diagnosis of DM2, Not having started TB treatment, Attend a selected health clinic, Sign a written informed consent

Exclusion Criteria:

* Unable to provide information, Pregnancy, HIV infection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Treatment success | Up to 6 months
  Bacteriological cure using sputum smear and culture
Blood glucose control | Up to 6 months
  mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Duadalupe Delgado Sanchez, PhD, Principal Investigator — Instituto Nacional de Salud Pública
Locations (1):
- Centro de Salud Camerino Mendoza, Orizaba, Veracruz, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez-Aguilar G, Serrano CJ, Castaneda-Delgado JE, Macias-Segura N, Hernandez-Delgadillo N, Enciso-Moreno L, Garcia de Lira Y, Valenzuela-Mendez E, Gandara-Jasso B, Correa-Chacon J, Bastian-Hernandez Y, Rodriguez-Moran M, Guerrero-Romero F, Enciso-Moreno JA. Associated Risk Factors for Latent Tuberculosis Infection in Subjects with Diabetes. Arch Med Res. 2015 Apr;46(3):221-7. doi: 10.1016/j.arcmed.2015.03.009. Epub 2015 Apr 10. PMID 25864989
- [Background] Riza AL, Pearson F, Ugarte-Gil C, Alisjahbana B, van de Vijver S, Panduru NM, Hill PC, Ruslami R, Moore D, Aarnoutse R, Critchley JA, van Crevel R. Clinical management of concurrent diabetes and tuberculosis and the implications for patient services. Lancet Diabetes Endocrinol. 2014 Sep;2(9):740-53. doi: 10.1016/S2213-8587(14)70110-X. PMID 25194887
- [Background] Delgado-Sanchez G, Garcia-Garcia L, Castellanos-Joya M, Cruz-Hervert P, Ferreyra-Reyes L, Ferreira-Guerrero E, Hernandez A, Ortega-Baeza VM, Montero-Campos R, Sulca JA, Martinez-Olivares Mde L, Mongua-Rodriguez N, Baez-Saldana R, Gonzalez-Roldan JF, Lopez-Gatell H, Ponce-de-Leon A, Sifuentes-Osornio J, Jimenez-Corona ME. Association of Pulmonary Tuberculosis and Diabetes in Mexico: Analysis of the National Tuberculosis Registry 2000-2012. PLoS One. 2015 Jun 15;10(6):e0129312. doi: 10.1371/journal.pone.0129312. eCollection 2015. PMID 26075393
- [Background] Ait-Khaled N, Enarson DA, Bencharif N, Boulahdib F, Camara LM, Dagli E, Djankine TK, Keita B, Karadag B, Ngoran K, Odhiambo J, Ottmani SE, Pham DL, Sow O, Yousser M, Zidouni N. Implementation of asthma guidelines in health centres of several developing countries. Int J Tuberc Lung Dis. 2006 Jan;10(1):104-9. PMID 16466046